CLINICAL TRIAL: NCT06322823
Title: A Pilot Study on Developing a One-step Direct Thawing Method on Human Blastocysts With Transcriptomic and Methylomic Comparison to Conventional Vitrified-thawing Method
Brief Title: Direct Thawing of Vitrified Human Blastocyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yiu Leung David Chan, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2010.432
Record Dates: First submitted 2024-03-13; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: IVF
MeSH Terms: interventions — Vitrification

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct thawing (Experimental)
  Interventions: Procedure: direct thawing
- commercially available vitrification thawing (Active Comparator)
  Interventions: Procedure: Vitrification

INTERVENTIONS:
Procedure: direct thawing — Vitrified blastocysts will be thawed directly into 1ml G-TL medium
  Arms: direct thawing
Procedure: Vitrification — Vitrified blastocysts will be thawed using commercially available one-step media.
  Arms: commercially available vitrification thawing

SUMMARY:
There are more than million frozen embryo transfers around the world each year; a faster, safer, and cheaper method can save a significant amount of money for patients undergoing IVF treatment worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to use direct-thawed blastocysts

Exclusion Criteria:

* Patients who are not willing to use direct-thawed blastocysts

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
blastocysts survival rate | up to 6 months
  The overall survival rate for thawed blastocysts using different thawing method will be compared.

SECONDARY OUTCOMES:
ferilization rate | up to 12 months
  The fertilization rate of frozen embryos using different thawing methods will be compared.
pregnancy rate | up to 12 months
  The pregnancy rate of patients who will be scheduled for the transfer of frozen embryos using different thawing methods will be compared.
live birth rate | up to 24 months
  The live birth rate of patients who will be scheduled for the transfer of frozen embryos using different thawing methods will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- David Yiu Leung Chan, Hong Kong, Hong Kong